CLINICAL TRIAL: NCT02284516
Title: A Phase 3, Multicenter, Randomized, Double-masked, and Placebo-controlled Study Evaluating the Efficacy and Safety of a 5.0% Concentration of Lifitegrast Ophthalmic Solution Compared to Placebo in Subjects With Dry Eye Disease and History of Recent Artificial Tear Use
Brief Title: A Study to Evaluate Efficacy and Safety of Lifitegrast in Subjects With Dry Eye (OPUS-3)
Acronym: OPUS-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHP606-304
Record Dates: First submitted 2014-10-30; First posted 2014-11-06 (Estimated); Results first posted 2017-03-15 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes | interventions — lifitegrast

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Lifitegrast (Experimental): Lifitegrast Ophthalmic Solution 5%, BID for 84 days
  Interventions: Drug: Lifitegrast
- Placebo (Placebo Comparator): Placebo to match active treatment, BID for 84 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lifitegrast — Lifitegrast Ophthalmic Solution 5%, BID for 84 days
  Arms: Lifitegrast
Drug: Placebo — Placebo to match active treatment, BID for 84 days
  Arms: Placebo

SUMMARY:
Evaluate the efficacy and safety of Lifitegrast in subjects with dry eye disease and a recent history of artificial tear use.

ELIGIBILITY:
Inclusion Criteria:

* Patient-reported history of Dry Eye Disease in both eyes.
* Use of over the counter artificial tears within the past 30 days.
* A negative urine pregnancy test for females and willingness to use adequate birth control throughout the study.
* Able and willing to comply with all study procedures.

Exclusion Criteria:

* Presence of an ocular condition that could affect the study parameters such as active ocular infections, ocular inflammation, glaucoma, or diabetic retinopathy;.
* Unwilling to stop wearing contact lenses during the study.
* LASIK or other ocular surgical procedures within 12 months prior to or during the study.
* Use of prohibited medications
* Significant medical conditions that could affect the study parameters.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 711 (Actual)
Dates: Start 2014-11-06 (Actual); Primary Completion 2015-10-05 (Actual); Study Completion 2015-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (41):
- United States (41):
  - University of Alabama at Birmingham, UAB School of Optometry, Birmingham, Alabama
  - Arizona Eye Center, Chandler, Arizona
  - Sall Research Medical Center, Artesia, California
  - United Medical Research Institute, Inglewood, California
  - North Valley Eye Medical Group, Inc, Mission Hills, California
  - Montebello Medical Eye Center, Inc., Montebello, California
  - Eye Research Foundation, Newport Beach, California
  - Arch Health Partners, Poway, California
  - Martel Eye Medical Group, Rancho Cordova, California
  - Shasta Eye Medical Group, Inc., Redding, California
  - West Coast Eye Care Associates, San Diego, California
  - Chicago Cornea Consultants, Ltd., Hoffman Estates, Illinois
  - Jackson Eye, SC, Lake Villa, Illinois
  - Price Vision Group, Indianapolis, Indiana
  - John-Kenyon American Eye Institute, New Albany, Indiana
  - Koffler Vision Group, Lexington, Kentucky
  - The Eye Care Institute, Louisville, Kentucky
  - Holpro Vision, Ltd., Union, Kentucky
  - Clinical Eye Research of Boston, Winchester, Massachusetts
  - Lifelong Vision Foundation, Chesterfield, Missouri
  - Tauber Eye Center, Kansas City, Missouri
  - Tekwani Vision Center, St Louis, Missouri
  - Ophthalmology Consultants, Ltd., St Louis, Missouri
  - Comprehensive Eye Care, Ltd., Washington, Missouri
  - Wellish Vision Institute, Las Vegas, Nevada
  - Abrams Eye Institute, Las Vegas, Nevada
  - Clinical Vision Research Center at SUNY, New York, New York
  - Ophthalmic Consultants Of Long Island, Rockville Centre, New York
  - South Shore Eye Care, LLP, Wantagh, New York
  - Abrams Eye Center, Cleveland, Ohio
  - Scott & Christie and Associates, PC, Cranberry Township, Pennsylvania
  - Matossian Eye Associates, Doylestown, Pennsylvania
  - Toyos Clinic, Nashville, Tennessee
  - The Cataract & Glaucoma Center, El Paso, Texas
  - Advanced Laser Vision and Surgical Institute, Houston, Texas
  - Whitsett Vision Group, Houston, Texas
  - University of Houston College of Optometry, Houston, Texas
  - The Eye Clinic of Texas (Houston Eye Associates), League City, Texas
  - Eye Clinics of South Texas, P.A., San Antonio, Texas
  - R and R Eye Research, LLC., San Antonio, Texas
  - See Clearly Vision, McLean, Virginia

REFERENCES:
- [Derived] Holland EJ, Jackson MA, Donnenfeld E, Piccolo R, Cohen A, Barabino S, Rolando M, Figueiredo FC. Efficacy of Lifitegrast Ophthalmic Solution, 5.0%, in Patients With Moderate to Severe Dry Eye Disease: A Post Hoc Analysis of 2 Randomized Clinical Trials. JAMA Ophthalmol. 2021 Nov 1;139(11):1200-1208. doi: 10.1001/jamaophthalmol.2021.3943. PMID 34617974
- [Derived] Holland EJ, Luchs J, Karpecki PM, Nichols KK, Jackson MA, Sall K, Tauber J, Roy M, Raychaudhuri A, Shojaei A. Lifitegrast for the Treatment of Dry Eye Disease: Results of a Phase III, Randomized, Double-Masked, Placebo-Controlled Trial (OPUS-3). Ophthalmology. 2017 Jan;124(1):53-60. doi: 10.1016/j.ophtha.2016.09.025. Epub 2016 Oct 27. PMID 28079022

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two participants from placebo arm (N=356) has taken study drug by mistake and considered for "Lifitegrast" arm (N=355). Therefore, Placebo (N=354), Lifitegrast (N=357) were considered for safety analysis.
Groups:
- Placebo: Placebo ophthalmic solution was administered to the ocular surface as a single eye drop twice daily in both eyes for 84 days.
- Lifitegrast: Lifitegrast 5% Ophthalmic Solution was administered to the ocular surface as a single eye drop twice daily in both eyes for 84 days.
Period: Overall Study
Arm/Group | Placebo | Lifitegrast
Started | 356 | 355
Safety Population | 354 (Two placebo participants were considered for Lifitegrast arm; Placebo safety analysis set (N= 354).) | 357 (Two placebo participants were included in Lifitegrast arm for safety analysis set (N=357).)
Completed | 318 | 319
Not Completed | 38 | 36

BASELINE CHARACTERISTICS:
Population: Randomized population included all participants screened for whom a randomization number was assigned.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Lifitegrast | Total
Number analyzed (Participants) | 356 | 355 | 711
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (14.84) | 58.8 (14.10) | 58.7 (14.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 269 | 268 | 537
  Male | 87 | 87 | 174

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Patient-Reported Eye Dryness Score to Day 84
Description: Eye dryness score was scored on a Visual Analogue Scale (VAS) ranges from 0-100 (0=no discomfort; 100=maximal discomfort).
Time Frame: Baseline to Day 84
Population: Intent to treat (ITT) population included all randomized participants who took at least 1 dose of investigational product with last observation carried forward (LOCF). Here, n = number of participants analyzed for the specific categories of each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Lifitegrast
Number analyzed (Participants) | 356 | 355
units on a scale
  Baseline (n=356, 355) | 69.0 (17.08) | 68.3 (16.88)
  Change from Baseline to Day 84 (n=353, 353) | -30.7 (28.01) | -37.9 (28.85)
Statistical Analysis 1: Comparison: Placebo vs Lifitegrast; Test type: Superiority or Other; p = 0.0007, ANOVA — The primary analysis was performed using a stratified 2-sample t-test (that is, analysis of variance [ANOVA]); Treatment Effect = 7.16, 95% CI 2-sided [3.04 to 11.28], Standard Error of Mean 2.096

2. Secondary Outcome: Change From Baseline in Patient-Reported Eye Dryness Score to Day 14 and Day 42
Description: as for outcome 1
Time Frame: Baseline to Day 14 and Day 42
Population: ITT population with LOCF. Here, n = number of participants analyzed for the specific categories of each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Lifitegrast
Number analyzed (Participants) | 356 | 355
units on a scale
  Baseline (n=356, 355) | 69.0 (17.08) | 68.3 (16.88)
  Change from Baseline to Day 14 (n=353, 352) | -15.0 (22.40) | -22.9 (25.44)
  Change from Baseline to Day 42 (n=353, 353) | -23.9 (25.99) | -33.2 (27.42)
Statistical Analysis 1: Comparison: Placebo vs Lifitegrast; Baseline and Day 14; Test type: Superiority or Other; p < 0.0001, ANOVA — The primary analysis was performed using a stratified 2-sample t-test (that is, analysis of variance [ANOVA]); Treatment Effect = 7.85, 95% CI 2-sided [4.33 to 11.37], Standard Error of Mean 1.792
Statistical Analysis 2: Comparison: Placebo vs Lifitegrast; Baseline and Day 42; Test type: Superiority or Other; p < 0.0001, ANOVA — The primary analysis was performed using a stratified 2-sample t-test (that is, analysis of variance [ANOVA]); Treatment Effect = 9.32, 95% CI 2-sided [5.44 to 13.20], Standard Error of Mean 1.976

ADVERSE EVENTS:
Time Frame: From start of the study drug administration upto Day 91 or Early termination (ET)
Description: Two participants from placebo arm (N=356) has taken study drug by mistake and considered for "Lifitegrast" arm (N=355). Therefore, Placebo (N=354), Lifitegrast (N=357) were considered for safety analysis.
Arm/Group | Placebo | Lifitegrast
Serious Adverse Events (participants affected / at risk) | 4/354 | 4/357
Other Adverse Events (participants affected / at risk) | 30/354 | 107/357
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=354) | Lifitegrast (N=357)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Lung neoplasm malignant (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Accelerated hypertension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=354) | Lifitegrast (N=357)
Instillation site irritation (General disorders) | 11 (12) | 65 (68)
Instillation site reaction (General disorders) | 19 (21) | 45 (51)
Dysgeusia (Nervous system disorders) | 1 (1) | 46 (46)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.